CLINICAL TRIAL: NCT01242020
Title: Microvascular Flow Assessment of the Periadventitial Adipose Tissue, Subcutaneous Adipose Tissue and Skeletal Muscle Using Contrast Enhanced Ultrasound (CEU); A Repeatability Study
Brief Title: Microvascular Flow Assessment Repeatability Study: The MARS Study
Acronym: MARS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to reliably reproduce, visualize, or quantify microvascular flow in the subcutaneous tissue, the skeletal muscle or peri-adventitia
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 811310
Record Dates: First submitted 2010-10-22; First posted 2010-11-16 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean Healthy Subjects (Other): "Lean" defined as (BMI ≥18 and ≤25)
  Interventions: Drug: Perflutren Lipid Microsphere Injectable Suspension
- Obese Healthy Subjects (Other): Obese grade I-II defined as (BMI>30 and ≤35)
  Interventions: Drug: Perflutren Lipid Microsphere Injectable Suspension

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere Injectable Suspension — 1.3 mL activated DEFINITY® diluted in 50 mL of preservative-free saline will be used

SUMMARY:
The purpose of this study is to test a method of imaging (taking a picture) of the abdomen (belly), neck, thigh and calf (lower leg) areas of the body, using ultrasound along with a drug which makes the pictures look clearer. Ultrasound is a type of imaging that uses sound waves to create a picture of the inside of the human body. Two sets of pictures will be taken on two different days to see if the results are the same each time.

DEFINITY® is a drug given intravenously (through the vein). DEFINITY® is approved by the FDA to be used as an ultrasound contrast agent (makes the pictures look clearer) while taking pictures of the heart. In this study, DEFINITY® will be used while taking pictures of blood vessels in your abdomen (belly), neck, thigh and calf (lower leg). Since this use of DEFINITY® is different than the use approved by the FDA, this study will be performed under an FDA Investigational New Drug (IND) application.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant/lactating women between the ages of 18 and 45;
2. Lean (BMI ≥18 and ≤25) or Obese grade I-II(BMI>30 and ≤35)
3. Provide written informed consent and sign HIPAA Waiver of Authorization
4. Be able and willing to follow all instructions and attend all study visits

Exclusion Criteria:

Subjects must not have been diagnosed with:

1. Coronary artery disease
2. Congestive heart failure
3. Congenital heart disease (Right-to-left, bi-directional, or transient right-to-left cardiac shunts)
4. Hypersensitivity to perflutren
5. Renal disease
6. Chronic obstructive pulmonary disease or Asthma
7. Primary or secondary pulmonary hypertension
8. Obstructive sleep apnea
9. Thyroid disease
10. Vasculitis
11. Peripheral arterial disease.
12. Cancer
13. Any type of immunosuppression
14. Any active infection (systemic or of the underlying skin or subcutaneous tissue).
15. Taking any prescribed medication for hypertension, dyslipidemia or diabetes.
16. Current or past smoking in the last 12 months.
17. Positive urine pregnancy test
18. Creatinine (Cr) above 1.4 mg/dl on screening evaluation
19. Hemoglobin (Hb) less than 10 mg/dl on screening evaluation
20. Aspartate Transaminase (AST) or Alanine Transaminase (ALT) two fold above upper limit of normal on screening evaluation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muredach P Reilly, MB, MSCE, Principal Investigator — University of Pennsylvania; Luis H. Eraso, MD, MPH, Study Director — University of Pennsylvania
Locations (1):
- Clinical and Translational Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lean Healthy Subjects | Obese Healthy Subjects
Started | 6 | 0
Completed | 3 | 0
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Failed screening | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lean Healthy Subjects | Obese Healthy Subjects | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Variability of Repeated Measures for Each Subject
Description: The variability of repeated measures for each subject, expressed as coefficient of variation (CV), in the periadventitial microvascular flow, subcutaneous microvascular flow and skeletal muscle flow.
Time Frame: up to 30 days
Population: Reliable data for periadventitial microvascular flow, subcutaneous microvascular flow, and skeletal microvascular flow were not collected for the Outcome Measure.
Arm/Group | Lean Healthy Subjects | Obese Healthy Subjects
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Microvascular Flow in the Periadventitial, Subcutaneous and Skeletal Muscle Tissues
Time Frame: up to 30 days
Population: Reliable data for periadventitial microvascular flow, subcutaneous microvascular flow, and skeletal muscle microvascular flow were not be collected for this outcome measure.
Arm/Group | Lean Healthy Subjects | Obese Healthy Subjects
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lean Healthy Subjects | Obese Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

LIMITATIONS AND CAVEATS:
Early termination (not feasible with available equipment) leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No